CLINICAL TRIAL: NCT05607550
Title: A Global, Phase 3, Randomized, Multicenter, Open-Label Study to Investigate the Efficacy and Safety of Furmonertinib Compared to Platinum-Based Chemotherapy as First-Line Treatment for Patients With Locally Advanced or Metastatic Non-Small Cell Lung Cancer (NSCLC) With Epidermal Growth Factor Receptor (EGFR) Exon 20 Insertion Mutations (FURVENT)
Brief Title: Study to Compare Furmonertinib to Platinum-Based Chemotherapy for Patients With Locally Advanced or Metastatic Non-Small Cell Lung Cancer (NSCLC) With Epidermal Growth Factor Receptor (EGFR) Exon 20 Insertion Mutations (FURVENT)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: ArriVent BioPharma, Inc. (Industry)
Collaborators: Allist Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FURMO-004; 2022-502977-41-00 (EU CTIS Number)
Record Dates: First submitted 2022-10-31; First posted 2022-11-07 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Metastatic Non-Small Cell Lung Cancer; Advanced Non-Small Cell Lung Cancer; EGFR Exon 20 Mutations
Keywords: Non-Small Cell Lung Cancer (NSCLC); Exon 20; Furmonertinib; Firmonertinib; AST2818; FURMO-004; Drug-Therapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — aflutinib; Platinum Compounds

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- furmonertinib 240 mg (Experimental)
  Interventions: Drug: furmonertinib 240 mg oral, daily
- furmonertinib 160 mg (Experimental)
  Interventions: Drug: furmonertinib 160 mg oral, daily
- platinum-based chemotherapy (Active Comparator): carboplatin or cisplatin based on investigator's choice + pemetrexed intravenously
  Interventions: Drug: platinum-based chemotherapy

INTERVENTIONS:
Drug: furmonertinib 240 mg oral, daily — furmonertinib tablet
  Other Names: AST2818
  Arms: furmonertinib 240 mg
Drug: furmonertinib 160 mg oral, daily — furmonertinib tablet
  Other Names: AST2818
  Arms: furmonertinib 160 mg
Drug: platinum-based chemotherapy — (carboplatin or cisplatin based on investigator's choice) + pemetrexed intravenously (IV)
  Arms: platinum-based chemotherapy

SUMMARY:
Global, Phase 3, randomized, multicenter, open-label study evaluating the efficacy and safety of furmonertinib (firmonertinib) at 2 dose levels (160 mg once daily [QD] and 240 mg QD) compared to platinum-based chemotherapy in previously untreated patients with locally advanced or metastatic non-squamous Non-Small Cell Lung Cancer (NSCLC) with Epidermal Growth Factor Receptor (EGFR) exon 20 insertion mutations. A target of approximately 375 patients will be randomized in a 1:1:1 ratio to treatment with furmonertinib 240 mg QD, furmonertinib 160 mg QD, or platinum-based chemotherapy.

ELIGIBILITY:
Key Inclusion Criteria:

* Histologically or cytologically documented, locally advanced or metastatic non-squamous Non-Small Cell Lung Cancer (NSCLC) not amenable to curative surgery or radiotherapy.
* Documented results of the presence of an Epidermal Growth Factor Receptor (EGFR) exon 20 insertion mutation in tumor tissue or blood from local or central testing.
* No prior systemic anticancer therapy regimens received for locally advanced or metastatic Non-Small Cell Lung Cancer (NSCLC) including prior treatment with any Epidermal Growth Factor Receptor (EGFR)-targeting agents (e.g., previous (EGFR) TKIs, monoclonal antibodies, or bispecific antibodies).
* Patients who have received prior neo-adjuvant and/or adjuvant chemotherapy, immunotherapy, or chemo radiotherapy for non-metastatic disease (excluding EGFR-TKIs) must have experienced a treatment free interval of at least 12 months.
* Patients with a history of treated CNS metastases or new asymptomatic CNS metastases are eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 398 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-08-15 (Estimated); Study Completion 2028-02-15 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) determined by blinded independent central review (BICR) | Up to 32 months after first dose

SECONDARY OUTCOMES:
Overall Survival (OS) | Up to 62 months after first dose
PFS determined by investigator assessment | Up to 36 months after first dose
Overall response rate (ORR) | Up to 36 months after first dose
Duration of response (DOR) | Up to 36 months after first dose
Time to second Progression Free Survival (PFS2) | Up to 36 months after first dose
PFS by blinded independent central review (BICR) in patients with a history or presence of brain metastases at baseline | Up to 36 months after first dose
Time to central nervous system (CNS) metastases by BICR | Randomization up to ≤30 days after last dose
CNS ORR evaluated by BICR | Randomization up to ≤30 days after last dose
CNS DOR evaluated by BICR | Randomization up to ≤30 days after last dose
CNS PFS evaluated by BICR | Randomization up to ≤30 days after last dose
Change in European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (QLQ-C30) | Randomization up to ≤30 days after last dose
  QLQ-C30 is a cancer-specific questionnaire comprised of 5 functional scales (physical, role, cognitive, emotional, and social functioning); 3 symptom scales (fatigue, pain, and nausea/vomiting); and a global health status/quality-of-life (QoL) scale. Six single-item scales are also included (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties).
Change in EORTC QLQ Lung Cancer Module Core 13 (QLQ LC13) | Randomization up to ≤30 days after last dose
  QLQ-LC13 is a cancer-specific questionnaire which comprises of 13 questions assessing lung cancer-associated symptoms (cough, hemoptysis, dyspnea, and site-specific pain), treatment-related side effects (sore mouth, dysphagia, peripheral neuropathy, and alopecia), and use of pain medication.
Change in Non-Small Cell Lung Cancer Symptom Assessment Questionnaire (NSCLC SAQ) | Randomization up to ≤30 days after last dose
  NSCLC-SAQ consists of 7 items assessing 5 NSCLC symptom concepts: cough, pain, dyspnea, fatigue, and poor appetite.
Number of incidence and severity of adverse events (AEs) as a measure of safety and tolerability of Furmonertinib | Up to 36 months after first dose
Plasma concentrations of furmonertinib and its major metabolite (AST5902) | Up to 36 months after first dose

CONTACTS AND LOCATIONS:
Overall Officials: Morgan Lam, Study Director — ArriVent BioPharm
Locations (196):
- United States (68):
  - Arrivent Investigative Site, Daphne, Alabama
  - Arrivent Investigative Site, Yuma, Arizona
  - Arrivent Investigative Site, Fayetteville, Arkansas
  - Arrivent Investigative Site, Beverly Hills, California
  - Arrivent Investigative Site, Fullerton, California
  - Arrivent Investigative Site, Long Beach, California
  - Arrivent Investigative Site, Los Alamitos, California
  - Arrivent Investigative Site, Napa, California
  - Arrivent Investigative Site, Orange, California
  - Arrivent Investigative site, Sacramento, California
  - Arrivent Investigative Site, San Diego, California
  - Arrivent Investigative Site, Santa Barbara, California
  - Arrivent Investigative Site, Santa Monica, California
  - Arrivent Investigative Site, Santa Rosa, California
  - Arrivent Investigative Site, Whittier, California
  - Arrivent Investigative Site, Hartford, Connecticut
  - Arrivent Investigative Site, Norwich, Connecticut
  - Arrivent Investigative Site, Fort Myers, Florida
  - Arrivent Investigative Site, St. Petersburg, Florida
  - Arrivent Investigative Site, The Villages, Florida
  - Arrivent Investigative Site, Peoria, Illinois
  - Arrivent Investigative Site, Rolling Meadows, Illinois
  - Arrivent Investigative Site, Fort Wayne, Indiana
  - Arrivent Investigative Site, Indianapolis, Indiana
  - Arrivent Investigative Site, South Bend, Indiana
  - Arrivent Investigative Site, Bethesda, Maryland
  - Arrivent Investigative Site, Frederick, Maryland
  - Arrivent Investigative Site, Rockville, Maryland
  - Arrivent Investigative Site, Fairhaven, Massachusetts
  - Arrivent Investigative Site, Lansing, Michigan
  - Arrivent Investigative Site, Bolivar, Missouri
  - Arrivent Investigative Site, Kansas City, Missouri
  - Arrivent Investigative Site, Saint Joseph, Missouri
  - Arrivent Investigative Site, St Louis, Missouri
  - Arrivent Investigative Site, Omaha, Nebraska
  - Arrivent Investigative Site, Belleville, New Jersey
  - Arrivent Investigative Site, Englewood, New Jersey
  - Arrivent Investigative Site, Florham Park, New Jersey
  - Arrivent Investigative Site, The Bronx, New York
  - Arrivent Investigative Site, Goldsboro, North Carolina
  - ArriVent Investigative Site, Pinehurst, North Carolina
  - Arrivent Investigative Site, Canton, Ohio
  - Arrivent Investigative Site, Cincinnati, Ohio
  - ArriVent Investigative Site, Cincinnati, Ohio
  - Arrivent Investigative Site, Cleveland, Ohio
  - Arrivent Investigative Site, Columbus, Ohio
  - Arrivent Investigative Site, Oklahoma City, Oklahoma
  - Arrivent Investigative Site, Tulsa, Oklahoma
  - Arrivent Investigative Site, Salem, Oregon
  - Arrivent Investigative Site, Gettysburg, Pennsylvania
  - ArriVent Investigative Site, Langhorne, Pennsylvania
  - Arrivent Investigative Site, York, Pennsylvania
  - Arrivent Investigative Site, Greenville, South Carolina
  - Arrivent Investigative Site, Sioux Falls, South Dakota
  - Arrivent Investigative Site, Memphis, Tennessee
  - ArriVent Investigative Site, Nashville, Tennessee
  - Arrivent Investigative Site, Abilene, Texas
  - ArriVent Investigative Site, Austin, Texas
  - Arrivent Investigative Site, Houston, Texas
  - Arrivent Investigative Site, Plano, Texas
  - Arrivent Investigative Site, Ogden, Utah
  - Arrivent Investigative Site, Salt Lake City, Utah
  - ArriVent Investigative Site, Fairfax, Virginia
  - Arrivent Investigative Site, Fredericksburg, Virginia
  - Arrivent Investigative Site, Bellingham, Washington
  - Arrivent Investigative Site, Spokane Valley, Washington
  - Arrivent Investigative Site, Tacoma, Washington
  - Arrivent Investigative Site, Appleton, Wisconsin
- Australia (4):
  - ArriVent Investigative Site, Heidelberg, Victoria
  - Arrivent Investigative Site, Blacktown
  - Arrivent Investigative Site, St Leonards
  - Arrivent Investigative Site, Woolloongabba
- Brazil (11):
  - ArriVent Investigative Site, Salvador, Estado de Bahia
  - ArriVent Investigative Site, Belo Horizonte, Minas Gerais
  - ArriVent Investigative Site, Rio de Janeiro, Rio de Janeiro
  - ArriVent Investigative Site, Pelotas, Rio Grande do Sul
  - ArriVent Investigative Site, Porto Alegre, Rio Grande
  - ArriVent Investigative Site, Blumenau, SC Cep
  - ArriVent Investigative Site, São José do Rio Preto, São Paulo
  - ArriVent Investigative Site, São Paulo, São Paulo
  - ArriVent Investigative Site, Liberdade, São Paulo/SP
  - ArriVent Investigative Site, Taubaté, Taubate SP
  - ArriVent Investigative Site, Porto Alegre
- Canada (2):
  - ArriVent Investigative Site, Edmonton, Alberta
  - ArriVent Investigative Site, Toronto, Ontario
- China (47):
  - Allist Investigative Site, Beijing, Beijing Municipality
  - Allist Investigative Site, Meizhou, Guangdong
  - Allist Investigative Site, Xuhui, Hai City
  - Allist Investigative Site, Hangzhou, Hangzhou
  - Allist Investigative Site, Cangzhou, Hebei
  - Allist Investigative Site, Shushan, Hefei
  - Allist Investigative Site, Zhengzhou, Henan
  - Allist Investigative Site, Changchun, Jilin
  - Allist Investigative Site, Weihai, Lingang Economic and Technological Development Zo
  - Allist Investigative Site, Nanning, Nanning
  - Allist Investigative Site, Yangpu, Shanghai Municipality
  - Allist Investigative Site, Xi’an, Shanxi
  - Allist Investigative Site, Taiyuan, Taiyuan
  - Allist Investigative Site, Kunming, Yunnan
  - Allist Investigative Site, Zhejiang, Zhejiang
  - Allist Investigative Site, Anyang
  - Allist Investigative Site, Changchun
  - Allist Investigative Site, Changsha
  - Allist Investigative Site, Chengdu
  - Allist Investigative Site, Chenzhou
  - Allist Investigative Site, Chongqing
  - Allist Investigative Site, Guangzhou
  - Allist Investigative Site, Harbin
  - Allist Investigative Site, Hefei
  - Allist Investigative Site, Huai'an
  - Allist Investigative Site, Huizhou
  - Allist Investigative Site, Jinan
  - Allist Investigative Site, Jining
  - Allist Investigative Site, Lanzhou
  - Allist Investigative Site, Lishui
  - Allist Investigative Site, Luoyang
  - Allist Investigative Site, Nanchang
  - Allist Investigative Site, Nanjing
  - Allist Investigative Site, Ningbo
  - Allist Investigative Site, Shanghai
  - Allist Investigative Site, Shantou
  - Allist Investigative Site, Shenyang
  - Allist Investigative Site, Shenzhen
  - Allist Investigative Site, Taiyuan
  - Allist Investigative Site, Tianjin
  - Allist Investigative Site, Weihui
  - Allist Investigative Site, Wuhan
  - Allist Investigative Site, Xiamen
  - Allist Investigative Site, Xianyang
  - Allist Investigative Site, Xinxiang
  - Allist Investigative Site, Xuzhou
  - Allist Investigative Site, Zhengzhou
- France (5):
  - Arrivent Investigative Site, Caen
  - Arrivent Investigative Site, Lyon
  - Arrivent Investigative Site, Marseille
  - Arrivent Investigative Site, Toulouse
  - Arrivent Investigative Site, Villejuif
- Israel (3):
  - ArriVent Investigative Site, Beersheba
  - ArriVent Investigative Site, Haifa
  - ArriVent Investigative Site, Jerusalem
- Italy (6):
  - ArriVent Investigative Site, Rozzano, Milan
  - ArriVent Investigative Site, Aviano, PN
  - ArriVent Investigative Site, Roma, Rome
  - ArriVent Investigative Site, Bari
  - Arrivent Investigative Site, Meldola
  - ArriVent Investigative Site, Milan
- Japan (13):
  - ArriVent Investigative Site, Kurume, Fukuoka
  - Arrivent Investigative Site, Akashi
  - Arrivent Investigative Site, Hirakata
  - Arrivent Investigative Site, Kashiwa
  - Arrivent Investigative Site, Nagoya
  - Arrivent Investigative Site, Ōsaka-sayama
  - Arrivent Investigative Site, Sapporo
  - Arrivent Investigative Site, Sendai
  - Arrivent Investigative Site, Shizuoka
  - Arrivent Investigative Site, Tokyo
  - ArriVent Investigative Site, Tokyo
  - Arrivent Investigative Site, Ube
  - Arrivent Investigative Site, Yokohama
- Malaysia (5):
  - ArriVent Investigative Site, George Town, Pulau Pinang
  - Arrivent Investigative Site, Cheras
  - Arrivent Investigative Site, Kota Bharu
  - Arrivent Investigative Site, Kuala Lumpur
  - Arrivent Investigative Site, Kuching
- Mexico (2):
  - ArriVent Investigative Site, Tuxtla Gutiérrez, Chiapas
  - ArriVent Investigative Site, Mexico City, Mexico City
- Netherlands (2):
  - Arrivent Investigative Site, Amsterdam
  - Arrivent Investigative Site, Harderwijk
- Philippines (4):
  - Arrivent Investigative Site, Cebu
  - Arrivent Investigative Site, Davao City
  - ArriVent Investigative Site, Manila
  - Arrivent Investigative Site, Pasig
- Singapore (2):
  - ArriVent Investigative Site, Singapore
  - Arrivent Investigative Site, Singapore
- South Korea (4):
  - ArriVent Investigative Site, Jungni I Gu, Seoul
  - Arrivent Investigative Site, Busan
  - Arrivent Investigative Site, Hwasun
  - Arrivent Investigative Site, Seoul
- Spain (5):
  - ArriVent Investigative Site, Málaga, Malaga
  - Arrivent Investigative Site, A Coruña
  - Arrivent Investigative Site, Barcelona
  - ArriVent Investigative Site, Madrid
  - Arrivent Investigative Site, Valencia
- Taiwan (6):
  - Arrivent Investigative Site, Chang-hua
  - Arrivent Investigative Site, Kaohsiung City
  - ArriVent Investigative Site, Kaohsiung City
  - ArriVent Investigative Site, Taichung
  - Arrivent Investigative Site, Tainan
  - Arrivent Investigative Site, Taipei
- Thailand (2):
  - Arrivent Investigative Site, Bangkok
  - Arrivent Investigative Site, Hat Yai
- United Kingdom (5):
  - ArriVent Investigative Site, Guildford, Surrey
  - Arrivent Investigative Site, Bebington, Wirral
  - ArriVent Investigative Site, London
  - ArriVent Investigative Site, Manchester
  - ArriVent Investigative Site, Sutton

IPD SHARING:
Plan to Share IPD: Undecided